CLINICAL TRIAL: NCT01178632
Title: A Double-blind, Randomized, Controlled, Phase III Study of an Herbal Medicine Association for Generalized Anxiety Disorder
Brief Title: Therapeutic Effect of an Herbal Medicine on Anxiety
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Millet Roux (Industry)
Responsible Party: FRANCISCO ALVES BORGES, MILLET ROUX
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MR4009
Record Dates: First submitted 2010-08-08; First posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Anxiety Disorders
Keywords: Herbal; Phytotherapy; Passiflora; Valeriana; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Valeriana extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Passiflora, Anxiety Disorders (Experimental): 1 tablet Passiflora;Crataegus;Salix; PO;BID
  Interventions: Drug: Passiflora
- Valeriane, Anxiety Disorder (Active Comparator): 1 tablet Valeriana officinalis, PO, BID
  Interventions: Drug: Valeriana officinalis

INTERVENTIONS:
Drug: Passiflora — 01 tablet Passiflora p.o., b.i.d.
  Other Names: PASSIFLORINE
  Arms: Passiflora, Anxiety Disorders
Drug: Valeriana officinalis — Active Comparator group will receive 01 tablet of Valeriana officinalis, p.o., b.i.d.
  Other Names: VALERIANE
  Arms: Valeriane, Anxiety Disorder

SUMMARY:
Phase III, double blind, randomized study, controlled by Valeriana officinalis L for evaluating the efficacy of association of Passiflora incarnata L; Crataegus Oxyacantha L and Salix alba L. in generalized anxiety disorder. The treatment period will last four weeks and be followed by a post treatment visit.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the clinical efficacy of the drug Passiflorine® (Passiflora incarnata L; Crataegus Oxyacantha L and Salix alba L) compared to Valeriana officinalis over a period of four weeks.

The improvement of anxiety disorders parameters (primary outcome) will be measured by the score of the Hamilton Anxiety Scale (HAM-A).

Does the administration of 2 tablets a day over a period of four weeks vs. Valeriana officinalis lead to an improvement in anxiety disorders?

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of generalized anxiety disorder
* HAM-A scale > 17 and <30

Exclusion Criteria:

* HAM-A scale > 30
* Psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-12 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Hamilton anxiety scale score | Four weeks
  The primary outcome measure for effectiveness will be the score of the Hamilton Anxiety Scale (HAM-A). This scale will be applied in the pre-treatment (baseline), in the two visits of the treatment and in the final visit (post-treatment). Tests will be done within groups, or between different assessments and baseline values, and intergroup comparisons, i.e. between the two treatment groups at each time.

SECONDARY OUTCOMES:
Insomnia gravity index | Four weeks
  The secondary outcome measure for effectiveness will be the score of the Insomnia gravity index. This questionnaire will be applied in the pre-treatment (baseline), in the two visits of the treatment and in the final visit (post-treatment). Tests will be done within groups, or between different assessments and baseline values, and intergroup comparisons, i.e. between the two treatment groups at each time.
Clinical global impression rate scale and Patient global evaluation rate scale | Four weeks
  The other secondary outcome measure for effectiveness will be the clinical global impression rate scale and patient global evaluation rate scale. These scales will be applied in the pre-treatment (baseline), in the two visits of the treatment and in the final visit (post-treatment). Tests will be done within groups, or between different assessments and baseline values, and intergroup comparisons, i.e. between the two treatment groups at each time.

CONTACTS AND LOCATIONS:
Overall Officials: MARIA ELISABETE A MORAES, MD, PhD, Study Director — CLINICAL PHARMACOLOGY UNIT - UNIFAC
Locations (1):
- Clinical Pharmacology Unit - Unifac, Fortaleza, Ceará, Brazil

REFERENCES:
- See also: ANXIETY DISORDERS — http://www.ncbi.nlm.nih.gov/pubmed
- See also: Passion Flower — http://www.ncbi.nlm.nih.gov/pubmed
- See also: Valeriana officinalis — http://www.ncbi.nlm.nih.gov/pubmed